CLINICAL TRIAL: NCT03811782
Title: Examining Conscious Motor Processing and the Effect of Single-task, Dual-task and Analogy Training on Walking During Rehabilitation by Older Adults at Risk of Falling in Hong Kong: A Randomized Controlled Trial
Brief Title: Effect of Single-task, Dual-task and Analogy Training During Gait Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Thomson Wai-Lung Wong, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW17-049
Record Dates: First submitted 2019-01-10; First posted 2019-01-22 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Fall; Balance; Reinvestment Propensity; Gait Rehabilitation
Keywords: conscious motor processing; single-task training; dual-task training; analogy training; gait rehabilitation; reinvestment propensity; balance; fear of falling; older adults; Hong Kong

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single-task Training Group (Experimental): Single-task walking group
  Interventions: Behavioral: Single-task Training
- Dual-task Training Group (Experimental): Dual-task walking group
  Interventions: Behavioral: Dual-task Training
- Analogy Training Group (Experimental): Analogy walking group
  Interventions: Behavioral: Analogy Training

INTERVENTIONS:
Behavioral: Single-task Training — In each training session, all groups will have warm-up (5 minutes), balance training (5 minutes), body transport training (5 minutes), body transport with hand manipulation training (5 minutes), walking training with various difficulties in a 10 meters walkway with Single-task Training instructions (20 minutes) and cool down (5 minutes).
  Arms: Single-task Training Group
Behavioral: Dual-task Training — In each training session, all groups will have warm-up (5 minutes), balance training (5 minutes), body transport training (5 minutes), body transport with hand manipulation training (5 minutes), walking training with various difficulties in a 10 meters walkway with Dual-task Training instructions (20 minutes) and cool down (5 minutes).
  Arms: Dual-task Training Group
Behavioral: Analogy Training — In each training session, all groups will have warm-up (5 minutes), balance training (5 minutes), body transport training (5 minutes), body transport with hand manipulation training (5 minutes), walking training with various difficulties in a 10 meters walkway with Analogy Training instructions (20 minutes) and cool down (5 minutes).
  Arms: Analogy Training Group

SUMMARY:
The study aims to examine the effect of single-task, dual-task and analogy training during gait rehabilitation on conscious motor processing propensity, balance, walking ability and fear of falling by older adults at risk of falling in Hong Kong. One-hundred and five healthy older adults will be recruited from elderly community centres in Hong Kong by convenience sampling. They will be randomly assigned into 3 groups (i.e., single-task walking group (active control group), dual-task walking group and analogy walking group). Participants in different groups will have training sessions (about 45 minutes each) three times per week for 4 weeks in a group of 5 participants. A total of 12 sessions will be completed by each participant. All training sessions will be conducted by experienced Hong Kong registered Physiotherapists. In each training session, all groups will have warm-up (5 minutes), balance training (5 minutes), body transport training (5 minutes), body transport with hand manipulation training (5 minutes), walking training with various difficulties in a 10 meters walkway with different instructions in different walking groups (20 minutes) and cool down (5 minutes). Participants in the different groups will receive different instructions during walking training. Well- developed single-task (explicit), dual-task and analogy instructions will be utilized in the single-task walking group, dual-task walking group and analogy walking group, respectively. Each participant will undergo assessment sessions (total 3 assessment sessions) before training at baseline (T0), just after completion of all training sessions (T1) and 6 months after completion of all training sessions (T2). In the baseline assessment, a structural questionnaire will be used to ask for demographics, detailed history of fall incident, detailed medical history, social history and social-economic status of the participants. A battery of assessments will be done to assess physical and cognitive abilities of the participants in all assessment sessions. Single-task walking ability, dual-task walking ability, functional gait and balance assessment, cognitive function, fearing of falling and propensity for conscious motor processing.

All participants will also be asked to record their number of falls prospectively at the time between T1 (completion of all training sessions) and T2 (6 months after completion of all training sessions) using a calendar. The number of falls within the 6-month follow- up period will then be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or above;
* No history of cerebral vascular disease, Parkinson's disease or other neurological deficit;
* Chinese version of the Mini-Mental State Examination (MMSE-C) (Folstein, Folstein, & McHuge, 1975; Chiu, Lee, Chung, & Kwong, 1994) total score of equal or more than 24;
* Able to walk independently indoor for at least 10 meters;
* Older adults with moderate to high risk of falling, as indicated by the score of less than 24 out of 28 in the Tinetti Balance Assessment Tool (Tinetti, 1986).

Exclusion Criteria:

* Any potential participant who cannot meet the inclusion criteria.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Baseline propensity for conscious motor processing | Before the start of training
  The Chinese version Movement Specific Reinvestment Scale (MSRS-C) (Masters et al., 2005; Wong et al., 2015a; Wong et al., 2015b). The MSRS-C includes two sub-scales: Conscious motor processing and Movement self-consciousness. The scores for both sub-scales ranges from 5-30. A higher score indicate a higher propensity for conscious motor processing.
Change from baseline propensity for conscious motor processing upon completion of training | Upon completion of 12 Training Sessions (4 weeks of training)
  The Chinese version Movement Specific Reinvestment Scale (MSRS-C) (Masters et al., 2005; Wong et al., 2015a; Wong et al., 2015b). The MSRS-C includes two sub-scales: Conscious motor processing and Movement self-consciousness. The scores for both sub-scales ranges from 5-30. A higher score indicate a higher propensity for conscious motor processing.
Change from baseline propensity for conscious motor processing at 6 months after the completion of training | 6 months after the completion of Training
  The Chinese version Movement Specific Reinvestment Scale (MSRS-C) (Masters et al., 2005; Wong et al., 2015a; Wong et al., 2015b). The MSRS-C includes two sub-scales: Conscious motor processing and Movement self-consciousness. The scores for both sub-scales ranges from 5-30. A higher score indicate a higher propensity for conscious motor processing.

SECONDARY OUTCOMES:
Baseline single-task walking ability | Before the start of training
  10 meters comfortable and fast walking speed (Bohannon, 1997)
Change from baseline single-task walking ability upon completion of training | Upon completion of 12 Training Sessions (4 weeks of training)
  10 meters comfortable and fast walking speed (Bohannon, 1997)
Change from baseline single-task walking ability at 6 months after the completion of training | 6 months after the completion of Training
  10 meters comfortable and fast walking speed (Bohannon, 1997)
Baseline dual-task walking ability | Before the start of training
  10 meters comfortable and fast walking speed with concurrent verbal or visual-spatial dual-tasks of auditory stroop task (Siu, Catena, Chou, van Donkelaar, & Woollacott, 2008) or clock test (Plummer-D'Amato, Altmann, Saracino, Fox, Behrman, & Marsiske, 2008)
Change from baseline dual-task walking ability upon completion of training | Upon completion of 12 Training Sessions (4 weeks of training)
  10 meters comfortable and fast walking speed with concurrent verbal or visual-spatial dual-tasks of auditory stroop task (Siu, Catena, Chou, van Donkelaar, & Woollacott, 2008) or clock test (Plummer-D'Amato, Altmann, Saracino, Fox, Behrman, & Marsiske, 2008)
Change from baseline dual-task walking ability at 6 months after the completion of training | 6 months after the completion of Training
  10 meters comfortable and fast walking speed with concurrent verbal or visual-spatial dual-tasks of auditory stroop task (Siu, Catena, Chou, van Donkelaar, & Woollacott, 2008) or clock test (Plummer-D'Amato, Altmann, Saracino, Fox, Behrman, & Marsiske, 2008)
Baseline Tinetti Balance Assessment Tool score | Before the start of training
  Tinetti Balance Assessment Tool (Tinetti, 1986).
Change from baseline Tinetti Balance Assessment Tool score upon completion of training | Upon completion of 12 Training Sessions (4 weeks of training)
  Tinetti Balance Assessment Tool (Tinetti, 1986)
Change from baseline Tinetti Balance Assessment Tool score at 6 months after the completion of training | 6 months after the completion of Training
  Tinetti Balance Assessment Tool (Tinetti, 1986)
Baseline Timed 'Up & Go' Tests time | Before the start of training
  Timed 'Up & Go' Tests (TU&G(Podsiadlo & Richardson, 1991)
Change from baseline Timed 'Up & Go' Tests time upon completion of training | Upon completion of 12 Training Sessions (4 weeks of training)
  Timed 'Up & Go' Tests (TU&G(Podsiadlo & Richardson, 1991)
Change from baseline Timed 'Up & Go' Tests time at 6 months after the completion of training | 6 months after the completion of Training
  Timed 'Up & Go' Tests (TU&G(Podsiadlo & Richardson, 1991)
Baseline Berg Balance Scale score | Before the start of training
  Berg Balance Scale (BBS) (Berg, Wood Dauphinee, Williams & Gayton, 1989)
Change from baseline Berg Balance Scale score upon completion of training | Upon completion of 12 Training Sessions (4 weeks of training)
  Berg Balance Scale (BBS) (Berg, Wood Dauphinee, Williams & Gayton, 1989)
Change from baseline Berg Balance Scale score at 6 months after the completion of training | 6 months after the completion of Training
  Berg Balance Scale (BBS) (Berg, Wood Dauphinee, Williams & Gayton, 1989)
Cognitive function | Before the start of training
  The Chinese version Mini-Mental State Examination (MMSE-C) (Folstein et al., 1975; Chiu et al., 1994). A mark of 24 or above out of 30 is required to meet the inclusion criteria.
Baseline fear of falling | Before the start of training
  Fall Efficacy Scale (FES-13) (Tinetti, Richman, & Powell L, 1990; Tinetti, Leon, Doucette & Parker, 1994; Hellström & Lindmark, 1999). The FES-13 score ranges from 16-64. A higher score indicates greater fear of falling.
Change from baseline fear of falling upon completion of training | Upon completion of 12 Training Sessions (4 weeks of training)
  Fall Efficacy Scale (FES-13) (Tinetti, Richman, & Powell L, 1990; Tinetti, Leon, Doucette & Parker, 1994; Hellström & Lindmark, 1999). The FES-13 score ranges from 16-64. A higher score indicates greater fear of falling.
Change from baseline fear of falling at 6 months after the completion of training | 6 months after the completion of Training
  Fall Efficacy Scale (FES-13) (Tinetti, Richman, & Powell L, 1990; Tinetti, Leon, Doucette & Parker, 1994; Hellström & Lindmark, 1999). The FES-13 score ranges from 16-64. A higher score indicates greater fear of falling.
Number of falls between T1 and T2 (post training to 6 months after completion of training) | 6 months after the completion of Training
  Record of the the number of falls prospectively at the time between T1 (completion of all training sessions) and T2 (6 months after completion of all training sessions) using a calendar.

CONTACTS AND LOCATIONS:
Overall Officials: Thomson Wai Lung WONG, Principal Investigator — The University of Hong Kong
Locations (1):
- The HKJC Building for Interdisciplinary Research, Hong Kong, Hong Kong